CLINICAL TRIAL: NCT00854919
Title: An Long Term Trial on Effectiveness and Safety of Atypical Antipsychotic Agents in Augmenting SSRI-Refractory Obsessive-Compulsive Disorder
Brief Title: Effectiveness and Safety of Atypical Antipsychotic Agents in Augmenting SSRI-Refractory Obsessive-Compulsive Disorder
Acronym: OCDDRUG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Osaka City University (Other)
Other Study IDs: 18591305
Record Dates: First submitted 2009-03-02; First posted 2009-03-03 (Estimated); Last update posted 2009-03-03 (Estimated); Status verified 2005-12

CONDITIONS: SSRI-Refractory Obsessive-Compulsive Disorder
Keywords: obsessive-compulsive disorder; augmentation treatment; SSRI-refractory
MeSH Terms: conditions — Obsessive-Compulsive Disorder

ARMS (3):
- CBT (Experimental): All subjects received cognitive-behavioral therapy (CBT) during the study period.
  Interventions: Behavioral: exposure response prevention
- 1 (Experimental): Drug; Paroxetine (30-50mg/D)or Fluvoxamine (150-250mg/D), 1-year administration
  Interventions: Drug: atypical antipsychotic drug; Behavioral: exposure response prevention
- 2 (Active Comparator): Either risperidone (1-5mg/D), olanzapine (1-5mg/D) or quetiapine (25-100mg/D) was added to ongoing SSRI, the combination trial was continued at least for half a year.
  Interventions: Drug: atypical antipsychotic drug; Behavioral: exposure response prevention

INTERVENTIONS:
Drug: atypical antipsychotic drug — For SSRI-refractory group, either atypical antipsychotic such as mean doses of RIS (3.1±1.9mg/day), of OLZ (5.1±3.2mg/day), and of QET (60.0±37.3mg/day) was added on ongoing SSRI(Paroxetine, Fluvoxamine).
  Arms: 1; 2
Behavioral: exposure response prevention — After at least 12 weeks from treatment initiation, cognitive-behavioral therapy (CBT) using exposure and response prevention was added with psychoeducational interventions and behavioral analysis.

SUMMARY:
Objective: Although atypical antipsychotic drugs (AAPDs) have been found effective in the augmentation of serotonin reuptake inhibitors (SRIs) for treatment-resistant obsessive-compulsive disorder (OCD) in short terms trials, there are few data on the effectiveness and safety of these agents in clinical settings over the long term.

Method: Subjects (n=46) who responded to selective SRIs (SSRIs) in an initial 12-week trial were continued on SRI-monotherapy plus cognitive-behavioral therapy (CBT) for one year. Subjects (n=44) who failed to respond to SSRIs were randomly assigned to one of 3 AAPDs such as risperidone and were consecutively treated using SSRI+AAPD combined with CBT for a year.

DETAILED DESCRIPTION:
More recently, second-generation atypical antipsychotic drugs (AAPD) that modulate both 5-HT and DA function, such as risperidone (RIS), olanzapine (OLZ) and quetiapine (QET), have been found effective in the augmentation of SSRIs for treatment-resistant OCD.

Nevertheless, the AAPDs have been associated with common and serious adverse effects, such as body weight (BW) gain and metabolic dysregulation. Metabolic dysregulation includes glucoregulatory dysfunction and dyslipidemia. Indeed, studies of some AAPD in SSRI-refractory OCD patients have similarly reported significant BW gain. AAPD-induced BW gain may influence patients' adherence to medication and places them at risk for a broad range of medical problems.

Most work on AAPDs in treatment-refractory OCD has been conducted in the form of short-term efficacy studies. There have been fewer studies of the effectiveness, safety, and tolerability of these agents in the context of a clinic where CBT is also provided, and where treatment is continued for a significant period of time. In the current effectiveness study, we sought to examine the response of SSRI-refractory patients to augmentation with AAPDs, comparing adverse events in such compared to a control group of SSRI responders.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or over
* Patients were diagnosed as having obsessive-compulsive disorder by the Structured Clinical Interview for DSM-IV Patient version (SCID-P)
* They received standardized treatment for at least 1 year at the OCD clinic in our university hospital.
* Each subject gave written informed consent to take part after receiving a complete description of this study.
* All subjects were free of medical illness based on results of physical examination and screening tests of blood and urine, and no subjects received any lipid lowering or hypoglycemic agent during the 1-year study period.

Exclusion Criteria:

* Current clinically significant medical conditions such as diabetes

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2006-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Yale-Brown Obsessive-Compulsive Scale | 1 year

SECONDARY OUTCOMES:
yale-Brown Obsessive-Compulsive Scale | 1 year
BMI, TG, T-CHO, FBS | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Neuropsychiatry, Osaka City University, graduate School of Medicine, Osaka, Osaka, Japan

REFERENCES:
- [Derived] Matsunaga H, Nagata T, Hayashida K, Ohya K, Kiriike N, Stein DJ. A long-term trial of the effectiveness and safety of atypical antipsychotic agents in augmenting SSRI-refractory obsessive-compulsive disorder. J Clin Psychiatry. 2009 Jun;70(6):863-8. doi: 10.4088/JCP.08m04369. Epub 2009 May 5. PMID 19422759